CLINICAL TRIAL: NCT00396357
Title: A Multicenter, Double-blind, Randomized Parallel-group, Study to Demonstrate the Effect of 24 Weeks Treatment With Vildagliptin 100 mg qd as add-on to Metformin 500 mg Bid Compared to Metformin 1000 mg Bid in Patients With Type 2 Diabetes Inadequately Controlled on Metformin 500 mg Bid Monotherapy
Brief Title: Efficacy/Safety of Vildagliptin and Metformin Combination Therapy in Patients With Type 2 Diabetes Not Well Controlled With Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23104
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; hemoglobin A1c; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- vildagliptin + metformin (Experimental)
  Interventions: Drug: Vildagliptin
- Metformin (Active Comparator)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: Vildagliptin
  Arms: vildagliptin + metformin
Drug: metformin
  Arms: Metformin

SUMMARY:
This study is designed to evaluate the efficacy and safety of vildagliptin in combination with metformin 500 mg bid compared to metformin 1000 mg bid in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 18-78 years inclusive
* Type 2 diabetes diagnosis at least 2 months prior to study entry
* Body mass index in the range of 22-45 kg/m2
* HbA1c in the range of 6.5 to 9% inclusive
* Fasting plasma glucose <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* A history of type 1 diabetes
* Evidence of significant diabetic complications
* Treatment with insulin or any other oral antidiabetic agents
* Congestive heart failure requiring pharmacologic treatment
* Clinically significant renal dysfunction defined by metformin labeling criteria (serum creatinine levels >/= 1.5 mg/dl (males) and >/= 1.4 mg/dl (females)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin A 1 c (HbA1c) after 24 weeks of treatment | 24 weeks

SECONDARY OUTCOMES:
Adverse event profile after 24 weeks of treatment | 24 weeks
Gastrointestinal tolerability after 24 weeks of treatment | 24 weeks
Patients with endpoint HbA1c <7% and <6.5% after 24 weeks | 24 weeks
Patients with reduction in HbA1c >0.7% after 24 weeks | 24 weeks
Change from baseline in fasting plasma glucose after 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Novartis Investigative Site, Multiple Locations, Germany

REFERENCES:
- See also: Results for CLAF237A23104 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2654